CLINICAL TRIAL: NCT00985179
Title: Promoting the Adoption and Maintenance of a Physically Active Lifestyle and a Nutrition Rich in Vitamins With the Help of Two Theory-based Computerized Interventions "BI Vit" (Boehringer Ingelheim for a Nutrition Rich in Vitamines) and "BI Active" (Boehringer Ingelheim for Physical Activity) for Employees
Brief Title: Increasing Vitamin Intake and Physical Activity
Acronym: BIV-BIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freie Universität Berlin (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sonia Lippke, Dr.; Assistant Professor (C1), Freie Universität Berlin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FU-19-4711-008; BI Vit; BI Activ
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2011-06

CONDITIONS: Heart Diseases; Diabetes Mellitus, Type 2; Behavior; Motivation
Keywords: Randomized Controlled Trial; evidence- and theory-based behavioral intervention; expert system; stages of change; motivational interviewing; tailoring; Self Care; Expert Systems
MeSH Terms: conditions — Heart Diseases; Diabetes Mellitus, Type 2; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (IG) (Experimental): Employees in the IG will receive an interactive, computerized expert system which tailors treatment components to the individual needs of them
  Interventions: Behavioral: Intervention Group (IG)
- Waiting control group (WCG) (No Intervention)

INTERVENTIONS:
Behavioral: Intervention Group (IG) — Employees in the IG will receive an interactive, computerized expert system which tailors treatment components to the individual needs of them
  Other Names: HAPA-based stage-matched intervention
  Arms: Intervention Group (IG)

SUMMARY:
To help employees to adopt and maintain a healthy lifestyle, it is imperative to increase their self-management competencies. Aim of this research project is to evaluate an evidence- and theory-based computerized expert system in comparison to waiting control group. Employees will be treated psychologically and followed up over 18 months. The computerized expert system is expected to help employees significantly changing their lifestyle. The intervention is hypothesized to improve self-management competencies over and above the regular check-up at their medical appointment (i.e., waiting control group).

DETAILED DESCRIPTION:
In a change setting (employees having a regular medical appointment), two interventions (one for nutrition change and one for activity change) will follow and assessments over a time period of 12 to 20 weeks will be conducted afterwards. Study participants in the intervention groups receive an interactive, computerized expert system (Intervention Group, IG). Individuals in the waiting control group (WCG) get nothing. Employees (N = 1000) will be recruited at their regular medical appointment. Study participants will be followed up over three measurement points: One to nine weeks after T1, T2 will take place. Five to 13 weeks after T1 the T3 measurement will be conducted.

The hypotheses are: In comparison to the WCG the employees in the IG are expected to have a higher motivation, to adopt a healthy lifestyle, to perform more health behavior and to be less likely to relapse into previous unhealthy routines. Also, IG employees will be healthier as well as they will report more quality of life, more work satisfaction and more occupational efficiency . In comparison to WCG, the IG is also hypothesized to be more effective than the WCG regarding social-cognitive predictors of behavior.

Moreover, the interventions are supposed to be more effective for individuals with more risk factors (obese ect.). After successful evaluation and some adoptions the intervention will be implemented as a self-help program in all eligible employees in the Intranet.

ELIGIBILITY:
Inclusion Criteria:

* to be capable of exercising on their own at a minimum level and/or to consume fruits and vegetables
* able to fill out a questionnaire (no illiteracy)
* adequate German language ability

Exclusion Criteria:

* no internet access
* no computer with keyboard

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
health behavior (physical activity & fruits and vegetables) | 13 weeks

SECONDARY OUTCOMES:
subjective health | 13 weeks
work satisfaction | 13 weeks
motivation/volition | 13 weeks
social-cognitive predictors of behavior (self-efficacy, action control etc.) | 13 weeks
objective health measures (body mass index, cholesterol, blood glucose ect.) | 13 weeks
perceived occupational efficiency | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ernsting, Principal Investigator — Freie Universitaet Berlin
Locations (1):
- Freie Universitaet Berlin, Berlin, State of Berlin, Germany